CLINICAL TRIAL: NCT02870517
Title: The Effect of Music on Pre-operative Stress in Pediatric Orthopedic Patients
Brief Title: Pre-operative Stress Reduction With Music
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Carolyn Barbieri, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005361
Record Dates: First submitted 2016-08-01; First posted 2016-08-17 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Pre-operative Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxing Music (Experimental): Participants will listen to relaxing music through noise-cancelling headphones during induction.
  Interventions: Other: Relaxing Music
- No Music (Active Comparator): Participants will wear noise-cancelling headphones during induction but no music will be played through them.
  Interventions: Other: No Music

INTERVENTIONS:
Other: Relaxing Music — Relaxing music, will be played through noise-cancelling headphones during induction of anesthesia. All of the songs used in this study will have <60 BPM, be instrumental rather than lyrical, and utilize predictable chord progressions. Music will be divided into several themed playlists which will be focused on the type of instruments involved including guitar, steel drum, and piano. The patient will listen to the music through noise-cancelling headphones beginning fifteen minutes prior to induction and ending one minute after intubation.
  Arms: Relaxing Music
Other: No Music — The patient will wear noise-cancelling headphones beginning fifteen minutes prior to induction and ending one minute after intubation.
  Arms: No Music

SUMMARY:
The purpose of this study is to assess the effect of music, played prior to a surgical procedure, on stress levels during induction of anesthesia. Hypothesis: playing "calming" music, pre-selected by the investigator and the patient, beginning just prior to induction and terminating after induction will positively reduce the patient's heart rate, blood pressure, and respiratory rate during this period. For this study, noise-cancelling headphones with the ability to play music via an iPod will be utilized.

DETAILED DESCRIPTION:
Reduced stress and relaxation positively contribute to patient healing after surgery (1). Reduction of stress associated with surgery is even more important in children, for whom a traumatic experience can have even more damaging and long-lasting effects (2). One stress-reduction technique of current interest is music. In global studies outside of the surgical realm, music has been shown to reduce heart rate, blood pressure, respiratory rate, and stress hormone levels as well as alleviate anxiety (3).

Evidence has also been found that listening to music pre-operatively in both adult and pediatric cases can reduce patients' stress and anxiety levels before surgery (3,7) Of the studies that have addressed the benefits of pre-operative music, however, none have assessed the impact of pre-operative music on stress levels during induction. In addition, almost all prior studies of the benefits of perioperative music have assessed the effect of only one style of music on each patient group. This set-up is beneficial in eliminating variables within the study design, but it fails to consider the individuality of each patient and what he/she might find to be relaxing. This study aims to assess the effect of music (selected by the pediatric patient from one of several pre-compiled playlists) played pre-operatively and during induction on patient stress levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 - 16 years
* Present to the OR for correction of an orthopedic complaint not involving the head or neck
* Consent to participate in the study obtained from both the guardian and child
* Patients and guardians are English-speaking

Exclusion Criteria:

* Hearing impairments or ear abnormalities
* Pre-existing issues with substance abuse, anxiety, or depression
* Pre-existing psychiatric disorders

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate from baseline recorded when the headphones are placed on the patient | 15 minutes after headphones are applied, at arrival in the operating room, during induction, during intubation, and one minute after intubation

SECONDARY OUTCOMES:
Change in Blood Pressure from baseline recorded when the headphones are placed on the patient | 15 minutes after headphones are applied, at arrival in the operating room, during induction, during intubation, and one minute after intubation
Change in Respiratory Rate from baseline recorded when the headphones are placed on the patient | 15 minutes after headphones are applied, at arrival in the operating room, during induction, during intubation, and one minute after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Barbieri, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holden-Lund C. Effects of relaxation with guided imagery on surgical stress and wound healing. Res Nurs Health. 1988 Aug;11(4):235-44. doi: 10.1002/nur.4770110405. PMID 3043570
- [Background] Oral R, Ramirez M, Coohey C, Nakada S, Walz A, Kuntz A, Benoit J, Peek-Asa C. Adverse childhood experiences and trauma informed care: the future of health care. Pediatr Res. 2016 Jan;79(1-2):227-33. doi: 10.1038/pr.2015.197. Epub 2015 Oct 13. PMID 26460523
- [Background] Daniel E. Music used as anti-anxiety intervention for patients during outpatient procedures: A review of the literature. Complement Ther Clin Pract. 2016 Feb;22:21-3. doi: 10.1016/j.ctcp.2015.11.007. Epub 2015 Dec 1. PMID 26850800
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695